CLINICAL TRIAL: NCT01640873
Title: A Randomized Double-Blind Placebo-Controlled Single and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-8655 in Subjects With Type 2 Diabetes
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-8655 in Participants With Type 2 Diabetes (MK-8655-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8655-002; MK-8655-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-8655 80 mg/MK-8655 320 mg (Experimental): Participants received a single dose of MK-8655, 80 mg on Day 1 and then MK-8655 320 mg, once daily, starting on Day 3 for 14 consecutive days.
  Interventions: Drug: MK-8655
- Placebo (Placebo Comparator): Participants received a single dose of placebo to MK-8655, 80 mg on Day 1 and then placebo to MK-8655 320 mg, once daily, starting on Day 3 for 14 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8655 — Participants will receive MK-8655 as a single dose on Day 1. Participants will receive MK-8655, once a day (q.d.), for 14 consecutive days (Day 3 through Day 16). MK-8655 doses may be adjusted downward based on the results of ongoing studies.
  Arms: MK-8655 80 mg/MK-8655 320 mg
Drug: Placebo — Participants will receive Placebo as a single dose on Day 1. Participants will receive Placebo, q.d., for 14 consecutive days (Day 3 through Day 16).
  Arms: Placebo

SUMMARY:
This study will assess the initial safety, tolerability, pharmacokinetics, and pharmacodynamics of MK-8655, after single and multiple daily oral administrations to participants with Type 2 Diabetes (T2DM). The study will assess the reduction in fasting plasma glucose concentrations from baseline after multiple daily administrations of MK-8655.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-child bearing potential
* Body Mass Index ≤40 kg/m^2
* Diagnosis of Type 2 Diabetes (T2DM) and is either drug naive or is being treated with metformin only
* In good health except for T2DM
* Willing to follow a standard diet
* Nonsmoker and/or no use of nicotine or nicotine-containing products for 6 months

Exclusion Criteria:

* Mentally or legally incapacitated
* History of stroke, chronic seizures, or major neurological disorder
* History of clinically significant endocrine (except T2DM), gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* History of neoplastic or myeloproliferative diseases
* Has clinical unstable or rapidly progressing diabetic retinopathy, neuropathy, and/or frequent nausea, bloating or vomiting, severe gastroesophageal reflux or early satiety
* Has a history of Type 1 Diabetes and/or history of ketoacidosis
* Use of any lipid-lowering therapies in the past 3 months
* Non-permitted medication for a co-morbid condition
* Excessive alcohol or caffeine use
* Participation in another investigational study within 4 weeks prior to this study
* A history of significant multiple and/or severe allergies or anaphylactic reactions
* Regular user of any illicit drugs or history of alcohol abuse within 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-09-19 (Actual); Primary Completion 2012-12-20 (Actual); Study Completion 2012-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant was a male or female (of non-child bearing potential) between 18 to 65 years of age with a diagnosis of Type 2 diabetes mellitus (T2DM) and was either drug naïve or was being treated with metformin only.
Period: Overall Study
Arm/Group | MK-8655 80 mg/MK-8655 320 mg | Placebo
Started | 22 | 11
Completed | 20 | 10
Not Completed | 2 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8655 80 mg/MK-8655 320 mg | Placebo | Total
Number analyzed (Participants) | 22 | 11 | 33
Age, Customized [Number; unit: Participants]
  31 to 63 years | 22 | 11 | 33
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All randomized participants
  Participants
    Female | 11 | 4 | 15
    Male | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Adverse Events
Description: An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 14 days after the last dose of study drug (Up to 31 days)
Population: All participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8655 80 mg/MK-8655 320 mg | Placebo
Number analyzed (Participants) | 22 | 11
Participants | 11 | 7

2. Primary Outcome: Number of Participants Discontinuing Study Drug Due to an Adverse Event
Description: as for outcome 1
Time Frame: Up to 17 days
Population: All participants who received at least one dose of the investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8655 80 mg/MK-8655 320 mg | Placebo
Number analyzed (Participants) | 22 | 11
Participants | 0 | 0

3. Primary Outcome: Fasting Plasma Glucose (FPG)
Description: Blood for fasting plasma glucose (central laboratory) was obtained after at least 10 hours overnight fast.
Time Frame: Day 16 (Predose)
Population: The analysis population was participants who complied with the protocol sufficiently to ensure that these data would likely exhibit the effects of treatment, according to the underlying scientific model. Compliance covered such considerations as exposure to treatment, availability of measurements and absence of major protocol violations.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MK-8655 80 mg/MK-8655 320 mg | Placebo
Number analyzed (Participants) | 22 | 11
mg/dL | 195.5 (52.5) | 211.8 (70.2)
Statistical Analysis 1: Comparison: MK-8655 80 mg/MK-8655 320 mg vs Placebo; Test type: Other; p = 0.356, Constrained longitudinal data analysis — The posterior probability that the reduction in FPG is ≥ 20 mg/dL is 0.06, and hence, the FPG hypothesis was not met; Least Squares Mean Difference = -8.50, 90% CI 2-sided [-47.4 to 30.4]

4. Secondary Outcome: True Geometric Mean Plasma Concentrations of MK-8655 After Single and Multiple Drug Doses at 24 Hours Post Dose (C24)
Description: C24hr was log transformed and analyzed based on a linear mixed effects model containing fixed effects for treatment, day and treatment by day interaction and a random effect for the participant.
Time Frame: 24 hours post dose on Days 1, 7, and 14
Population: The analysis population was participants who complied with the protocol sufficiently to ensure that these data would likely exhibit the effects of treatment, according to the underlying scientific model. No pharmacokinetic analysis for C24 was performed for participants receiving placebo.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: uM
Arm/Group | MK-8655 80 mg/MK-8655 320 mg | Placebo
Number analyzed (Participants) | 22 | 0
uM
  Day 1, MK-8655 80 mg, single dose | 0.133 (68.2) |
  Day 1, MK-8655 320 mg, multiple doses | 0.477 (72.1) |
  Day 7, MK-8655 320 mg, multiple doses | 0.549 (66.9) |
  Day 14, MK-8655 320 mg, multiple doses | 0.612 (69.4) |

5. Secondary Outcome: 24-Hour Weighted Mean Glucose (WMG)
Description: The WMG provides an integrated assessment of the glycemic exposure over the 24-hour period. To reduce variability of the baseline (before any study drug administration) WMG, participants were domiciled in the test facility at least 36 hours prior to Day 1, where standard meals were provided, and physical activity was monitored. The WMG was derived from multiple glucose values collected during both fasting and post-meal periods. The sample scheme for the 18 point glucose measurements used in this study had many samples taken in the very early morning hours, as well as the first three hours after meals. WMG was calculated as the area under the curve (AUC) of the glucose concentrations divided by the duration of time of samples collected.
Time Frame: Day 15: Predose, 2, 3, 4, 5, 6, 7, 8, 9, 11, 12, 13, 14, 15, 16, 18, 21, 23 hours post-dose.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MK-8655 80 mg/MK-8655 320 mg | Placebo
Number analyzed (Participants) | 22 | 11
mg/dL | 205.5 (33.95) | 199.9 (78.81)
Statistical Analysis 1: Comparison: MK-8655 80 mg/MK-8655 320 mg vs Placebo; Test type: Other; p = 0.2714, Constrained longitudinal data analysis — The posterior probability that the reduction in 24h-WMG is ≥ 20 mg/dL is < 0.01, and hence, the 24h- WMG hypothesis was not met; Geometric Mean Ratio = 1.05, 90% CI 2-sided [0.92 to 1.19]

6. Secondary Outcome: Change From Baseline at 2 Hours Oral Glucose Tolerance Test
Description: Plasma glucose excursion was assessed during an oral glucose tolerance test (oGTT) following a single dose administration of MK-8655 in participants with T2DM.
Time Frame: Baseline and 2 hours after dosing on Days 1, 3, and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MK-8655 80 mg/MK-8655 320 mg | Placebo
Number analyzed (Participants) | 22 | 11
mg/dL
  Day 1 | 164.0 (41.4) | 134.7 (74.5)
  Day 3 | 162.3 (37.0) | 135.0 (74.1)
  Day 16: number analyzed (Participants) | 18 | 9
  Day 16 | 172.4 (39.2) | 156.1 (79.4)
Statistical Analysis 1: Comparison: MK-8655 80 mg/MK-8655 320 mg vs Placebo; Test type: Other — Day 1; p = 0.060, ANOVA; Placebo-corrected (MK-8655 / placebo); Geometric Mean Ratio = 1.22, 95% CI 2-sided [0.99 to 1.55]
Statistical Analysis 2: Comparison: MK-8655 80 mg/MK-8655 320 mg vs Placebo; Test type: Other — Day 3; p = 0.065, ANOVA; Placebo-corrected (MK-8655 / placebo); Geometric mean Ratio = 1.20, 95% CI 2-sided [0.98 to 1.47]
Statistical Analysis 3: Comparison: MK-8655 80 mg/MK-8655 320 mg vs Placebo; Test type: Other — Day 16; p = 0.217, ANOVA; Placebo-corrected (MK-8655 / placebo); Geometric Mean Ratio = 1.10, 95% CI 2-sided [0.89 to 1.37]

ADVERSE EVENTS:
Time Frame: Up to 31 days
Description: The analysis population was all participants who received at least one dose of the investigational drug.
Arm/Group | MK-8655 80 mg/MK-8655 320 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/11
Other Adverse Events (participants affected / at risk) | 11/22 | 7/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8655 80 mg/MK-8655 320 mg (N=22) | Placebo (N=11)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Tiredness (General disorders) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3)
Abrasion NOS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ferritin decreased (Investigations) | 1 (1) | 1 (1)
Glucose increased (Investigations) | 2 (2) | 1 (3)
Hypoglycaemic reaction (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.